CLINICAL TRIAL: NCT04697472
Title: Clinical Assessment of Upper Extremity Performance in Individuals With Spinal Cord Injury Using the LIFT System to Deliver Non-invasive Electrical Spinal Stimulation (ARC Therapy)
Brief Title: The Up-LIFT Study of Non-Invasive ARC Therapy for Spinal Cord Injury
Acronym: Up-LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ONWARD Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DOC1622; Pro00046320 (Other: Advarra)
Record Dates: First submitted 2020-12-04; First posted 2021-01-06 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Chronic Spinal Cord Injury
Keywords: SCI; Tetraplegia; ARC Therapy
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Functional task practice (FTP) followed by FTP + ARC Therapy (Experimental): Clinic-based functional task practice (FTP) for two months followed by FTP + ARC Therapy for an additional 2 months.
  Interventions: Device: LIFT System

INTERVENTIONS:
Device: LIFT System — The LIFT System delivers the ARC Therapy to improve upper extremity function in individuals with tetraplegia.

SUMMARY:
The Up-LIFT Study is a prospective, single-arm study designed to evaluate the safety and effectiveness of non-invasive electrical spinal cord stimulation (ARC Therapy) administered by the LIFT System to treat upper extremity functional deficits in people with chronic tetraplegia.

DETAILED DESCRIPTION:
The primary endpoint of this pivotal study will report device related safety and changes in established metrics of upper extremity performance after treatment with the study device.

To ensure that the benefits realized in the study are directly attributable to the ARC Therapy, all enrolled subjects will first undergo a guided, in-clinic conventional functional task practice (FTP) program lasting approximately two months to regain their upper extremity (UE) function. Performance gains realized during this wash-in period provide a subject specific control that reflects the limits of conventional functional task practice without stimulation (standard of care). At the conclusion of the wash-in period, subjects will complete pre-stimulation testing of UE function.

To test the additive benefit of training with stimulation, combined functional task practice and ARC Therapy will then be administered over a period of approximately two months using the LIFT System. Functional task practice will follow established rehabilitation protocols that are specific to the individual subject's specific needs and capabilities (Beekhuizen & Field-Fote, Functional Task Practice versus Functional Task Practice with Stimulation: Effects on Upper Extremity Function and Cortical Plasticity in Individuals with Incomplete Cervical Spinal Cord Injury, 2005). Training will be graded to accommodate performance improvement over time, thus maximizing the potential benefit to subjects. Subjects will participate in up to 20 in-clinic training sessions per month. At the end of training period, the improvement in UE function will be measured and used to assess the progress of primary study endpoints.

The choice of primary outcome measures for this pivotal study is dictated by the following factors -

1. Safety,
2. Relevance to UE function,
3. Capture improvements in performance, and
4. Magnitude of changes that are clinically meaningful.

All performance metrics will be assessed at enrollment, at the completion of the wash-in period and at the end of the ARC Therapy assessment period. Subjects with clinically meaningful gains in multiple performance domains resulting from the ARC Therapy with LIFT will be considered responders. Additionally, gains during the wash-in (control) period will be compared to gains during the ARC Therapy with LIFT (test) period. Safety will be evaluated throughout the entire study through periodic monitoring and analysis of all reported adverse events.

ELIGIBILITY:
Key Inclusion Criteria:

Subjects must meet all the following criteria:

1. At least 22 years old and no older than 75 years old at the time of enrollment
2. Non-progressive cervical spinal cord injury from C2-C8 inclusive
3. American Spinal Injury Association (ASIA) Impairment Scale (AIS) classification B, C, or D
4. Indicated for upper extremity training procedures by subject's treating physician or a physical therapist
5. Minimum 12 months post-injury
6. Capable of providing informed consent

Key Exclusion Criteria:

Subjects must not meet any of the following criteria:

1. Has uncontrolled cardiopulmonary disease or cardiac symptoms as determined by the Investigator
2. Has any unstable or significant medical condition that is likely to interfere with study procedures or likely to confound study endpoint evaluations like severe neuropathic pain, depression, mood disorders or other cognitive disorders
3. Has been diagnosed with autonomic dysreflexia that is severe, unstable, and uncontrolled
4. Requires ventilator support
5. Has an autoimmune etiology of spinal cord dysfunction/injury
6. Spasms that limit the ability of the subjects to participate in the study training as determined by the Investigator
7. Breakdown in skin area that will come into contact with electrodes
8. Has any active implanted medical device
9. Pregnant, planning to become pregnant or currently breastfeeding
10. Concurrent participation in another drug or device trial that may interfere with this study
11. In the opinion of the investigators, the study is not safe or appropriate for the participant

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events (SAEs) | Through completion of the study, an average of 16 months
  Safety demonstrated through observational data regarding the incidence of serious adverse events (SAEs) related to the use of the study device and treatment procedures will be reported.
Number of participants with change in upper extremity strength and function | Through completion of the study, an average of 16 months
  Change in upper extremity strength and function performance metrics after treatment with ARC Therapy administered by the LIFT System and Functional Task Practice (FTP) is assessed using ISNCSCI, GRASSP,CUE-T, pinch/grasp forces.
  The primary effectiveness outcome measure will test the hypothesis that a majority of the subjects will experience clinically significant improvement in UE performance metrics (defined as therapy responders) after treatment with ARC Therapy administered by the LIFT System and Functional Task Practice (FTP).

SECONDARY OUTCOMES:
Superiority of combined FTP and ARC Therapy with LIFT vs. FTP alone. | Through completion of the study, an average of 16 months
  Superiority as demonstrated by statistically significant difference in the proportion of subjects reporting improvement between the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Edelle Field-Fote, PT, PhD, Principal Investigator — Shepherd Center - Crawford Research Institute; Chet Moritz, PhD, Principal Investigator — University of Washington
Locations (14):
- United States (9):
  - Craig Hospital, Englewood, Colorado
  - Miller School of Medicine, The Miami Project to Cure Paralysis, Miami, Florida
  - Shepherd Center- Crawford Research Institute, Atlanta, Georgia
  - INSPIRE Laboratory, Spaulding Hospital, Cambridge, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - James J. Peters VA Medical Center, The Bronx, New York
  - Thomas Jefferson University/Magee Rehabilitation Hospitals, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington
- Canada (2):
  - International Collaboration on Repair Discoveries (ICORD), University of British Columbia, Vancouver, British Columbia
  - KITE Research Institute /University Health Network, Toronto, Ontario
- Netherlands (2):
  - Sint Maartenskliniek, Department of Rehabilitation, Nijmegen, Gelderland
  - Reade, Centre for Rehabilitation and Rheumatology, Amsterdam, North Holland
- Queen Elizabeth National Spinal Injuries Unit, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inanici F, Samejima S, Gad P, Edgerton VR, Hofstetter CP, Moritz CT. Transcutaneous Electrical Spinal Stimulation Promotes Long-Term Recovery of Upper Extremity Function in Chronic Tetraplegia. IEEE Trans Neural Syst Rehabil Eng. 2018 Jun;26(6):1272-1278. doi: 10.1109/TNSRE.2018.2834339. PMID 29877852
- [Background] Hoffman L, Field-Fote E. Effects of practice combined with somatosensory or motor stimulation on hand function in persons with spinal cord injury. Top Spinal Cord Inj Rehabil. 2013 Fall;19(4):288-99. doi: 10.1310/sci1904-288. PMID 24244094
- [Derived] Moritz C, Field-Fote EC, Tefertiller C, van Nes I, Trumbower R, Kalsi-Ryan S, Purcell M, Janssen TWJ, Krassioukov A, Morse LR, Zhao KD, Guest J, Marino RJ, Murray LM, Wecht JM, Rieger M, Pradarelli J, Turner A, D'Amico J, Squair JW, Courtine G. Non-invasive spinal cord electrical stimulation for arm and hand function in chronic tetraplegia: a safety and efficacy trial. Nat Med. 2024 May;30(5):1276-1283. doi: 10.1038/s41591-024-02940-9. Epub 2024 May 20. PMID 38769431